CLINICAL TRIAL: NCT00355043
Title: Efficacy of Zinc in the Treatment of Bronchiolitis and Prevention of Wheezing Respiratory Illness in Children Less Than Two Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, International Centre for Diarrhoeal Disease Resarch, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-027
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2006-07

CONDITIONS: Bronchiolitis
Keywords: Zinc treatment; Bronchiolitis; Wheezing; Children aged 2 months to 23 months; Diagnosed case of acute bronchiolitis
MeSH Terms: conditions — Bronchiolitis; Respiratory Sounds | interventions — Zinc Sulfate

INTERVENTIONS:
Drug: Zinc sulphate 20 mg

SUMMARY:
1. Bronchiolitis is a leading cause of morbidity and mortality in children. It is an acute, infectious illness of the lower respiratory tract resulting in obstruction of the bronchioles. The etiology is viral in the majority of the cases and RSV is the most commonly isolated agent. The disease is more common in younger children under 2 years of age. Children often receive unnecessary antibiotics and often require hospitalization. An episode of bronchiolitis can be followed by recurrent wheezing episodes. RSV bronchiolitis in the first year of life is one of the most important risk factors for the subsequent development of asthma in both developed and developing countries. Thus, bronchiolitis is a global public health problem. Zinc supplementation has been shown to be effective in both preventing and treating pneumonia. However, no study has particularly examined the effect of zinc on ARI associated with wheezing. This study aims to investigate whether zinc (20 mg/day) reduces1. the duration of bronchiolitis in children.2. the severity of bronchiolitis in children.3. the rate of hospitalization for bronchiolitis.3. future episodes of wheezing in children.

ELIGIBILITY:
Inclusion Criteria:

Children 2 months to 23 months old at the time of clinical diagnosis· Episode of wheezing for the first time Written consent· Who do not require hospitalization at the time of diagnosis

Exclusion Criteria:

History of asthma Chronic cardiac or respiratory disease (e.g.cyanotic heart disease -ASD) History of previous wheezing or bronchodilator therapy Gestational age at birth <34 weeks Suspected tuberculosis, active measles Any illness (severe malnutrition, sepsis, meningitis) that requires hospitalisation Who had zinc/placebo supplements during this study· H/o zinc intake within last 3 months· Whose caretakers withhold consent

Ages: 2 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Effect of zinc on the duration of bronchiolitis in children

SECONDARY OUTCOMES:
Effect of Zinc
The severity of bronchiolitis.
The rate of hospitalization.
Future episodes of wheezing.

CONTACTS AND LOCATIONS:
Overall Officials: Dilruba Nasrin, MBBS,PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh